CLINICAL TRIAL: NCT00553995
Title: Effect of Physical Inactivity on Endothelial Function
Brief Title: Effect of Salsalate on Bed Rest-Induced Vascular Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Principal Investigator, Naomi M Hamburg, Principal Investigator, Boston University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-23068
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — salicylsalicylic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salsalate (Experimental): Salsalate
  Interventions: Drug: salsalate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: salsalate — Salsalate 3-4 grams per day as tolerated for nine days
  Arms: Salsalate
Drug: Placebo
  Arms: Placebo

SUMMARY:
Physical inactivity induces vascular dysfunction and glucose intolerance during five days of bed rest. This study will investigate the effects of salsalate on these responses. Subjects will be randomized to treatment with salsalate or placebo for four days prior to initiation of bed rest. Vascular function in the brachial artery will be determined by ultrasound prior to treatment and before and after the 5-day bed rest protocol. We hypothesize that treatment with salsalate will be associated with protection again the development of glucose intolerance and vascular dysfunction in this setting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Pregnancy
* History of Coronary Artery Disease
* Diabetes Mellitus
* Hypertension
* Cigarette smoking
* History or family history of deep vein thrombosis or pulmonary embolism
* Abnormal renal function
* Liver function tests greater than two times the upper limit of normal
* Anemia
* Use of viagra or other PDE5 inhibitor
* Hypercholesterolemia
* Aspirin allergy/sensitivity
* Asthma with nasal polyps
* Peptic ulcer disease/Gastrointestinal bleeding
* Any ongoing drug treatment

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-05 (Actual); Primary Completion 2013-12-01 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
Reactive hyperemia in the femoral artery | 5 days

SECONDARY OUTCOMES:
Reactive hyperemia in the brachial artery | 5 days
Oral glucose tolerance test | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Hamburg, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University School of Medicine, Boston, Massachusetts, United States